CLINICAL TRIAL: NCT01722721
Title: Physicians Work Distribution in a Danish Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, assistant professor, University of Southern Denmark
Other Study IDs: SLB-ED-01-2012
Record Dates: First submitted 2012-10-24; First posted 2012-11-07 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Time Usage of ED Physicians

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
physicians in the Emergency Department spend their time on interviewing and examining patients, file documentation, communication with colleagues about the patients.

Introduction of IT technology aims to reduce the administrative workload. However it is the impression that more and more time are used behind the PC rather than at the side of the patient.

The aim of this study is to describe how the time is distributed between different task for an ED physician, and to analyse whether there are differences in time distribution if the physician is working in the outpatient area versus admission area of the ED.

ELIGIBILITY:
Inclusion Criteria:

ED physicians employed in the ED department

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Department physicians
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
time in minutes used by Emergency Department (ED) physician on direct patient contact, documentation, communication about the patient. | first 24 hours after patient arrival to ED
  the time measured in minutes used by the emergency physician on direct patient contact, examination and treatment, documentation in IT systems and communication with other health staff about the patient is counted by indepedent observer

REFERENCES:
- [Derived] Fuchtbauer LM, Norgaard B, Mogensen CB. Emergency department physicians spend only 25% of their working time on direct patient care. Dan Med J. 2013 Jan;60(1):A4558. PMID 23340186